CLINICAL TRIAL: NCT06294041
Title: A Pilot Randomised Control Trial of Sleep Restriction Therapy Versus Sleep Hygiene Education for Newly Diagnosed Breast Cancer Patients With Acute Insomnia
Brief Title: INvestigating the Value of Early Sleep Therapy
Acronym: INVEST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Strathclyde (Other)
Collaborators: University of Oxford (Other); University of Glasgow (Other); NHS Greater Glasgow and Clyde (Other); NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UEC23/52
Record Dates: First submitted 2024-02-15; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Acute Insomnia (Disorder)
Keywords: acute insomnia; breast cancer; prehabilitation; sleep restriction therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the SRT intervention, the research nurse, patients and most of the study team cannot be blinded to treatment allocation. However, the statistician will be blinded to treatment allocation (i.e., SRT or SHE) until after analysis is complete
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Restriction Therapy (SRT) (Other)
  Interventions: Behavioral: Sleep Restriction Therapy (SRT)
- Sleep Hygiene Education (Other)
  Interventions: Behavioral: Sleep Hygiene Education (SHE)

INTERVENTIONS:
Behavioral: Sleep Restriction Therapy (SRT) — SRT is a manualised, adaptive, behavioural insomnia intervention that is a key active ingredient within multi-component CBT-I. Our SRT protocol involves standardising and (where required) limiting a patient's time in bed with the aim of increasing homeostatic sleep pressure, over-riding cognitive and physiological arousal, and strengthening circadian control of sleep. Those randomised to the SRT arm will receive two online sessions supported by two telephone calls over a 4-week intervention phase. The intervention will be delivered by trained research nurses
  Arms: Sleep Restriction Therapy (SRT)
Behavioral: Sleep Hygiene Education (SHE) — SHE will be delivered via a booklet that provides information about lifestyle changes (e.g., reducing exercise in the evening, light snack before bedtime, reducing caffeine) and changes to the bedroom environment (e.g., dark room, comfortable mattress, optimal room temperature). Patients in the SHE condition will be instructed to implement the SHE advice over a 4-week period. One week after randomisation to SHE, the RA will telephone patients to check they understand the SHE advice and answer any questions they may have. SHE has successfully been used as a control condition in other trials evaluating SRT and does not have any therapeutic benefit for individuals with insomnia but is often part of usual care, so is a credible alternative to SRT.
  Arms: Sleep Hygiene Education

SUMMARY:
Twenty percent of breast cancer survivors have insomnia, which is defined as persistent trouble falling and/or staying asleep that results in difficulty functioning during the day. Sleep difficulties often begin at cancer diagnosis, become worse during cancer treatment, and continue into cancer survivorship. Insomnia interferes with daily activities and may cause other mental and physical health problems. It also makes it more difficult to cope with cancer treatment and makes recovery more challenging. For these reasons, it is important to address early signs of sleep problems in cancer patients by offering interventions that may prevent the development of insomnia.

Sleep Restriction Therapy is one such intervention, which helps improve night-time sleep by stabilising sleep patterns and reducing time spent in bed awake. Sleep Restriction Therapy has been used successfully to treat chronic insomnia in breast cancer survivors who have completed cancer treatment. However, it has never been tested on newly diagnosed breast cancer patients with early signs of sleep disturbance, who are undergoing cancer treatment.

This study will address this knowledge gap by randomly assigning newly diagnosed patients with poor sleep to receive either Sleep Restriction Therapy or a sleep hygiene education (SHE) control intervention. The study will assess sleep and mental health before and after both interventions to determine how feasible and acceptable Sleep Restriction Therapy is to patients and to plan for a future, larger study. Throughout, the investigators will work with patients with lived experience of breast cancer and poor sleep to ensure our study is informed by their expertise.

DETAILED DESCRIPTION:
The primary aim of this project is to assess the feasibility and inform the design of a full-scale RCT of SRT for newly diagnosed breast cancer patients with acute insomnia. Secondary aims of this project are to assess the effects of SRT alongside a sleep hygiene education (SHE) control on sleep, rest-activity rhythms, and mental health.

Participants will be recruited from breast cancer results clinics in two study sites. Our target population is newly diagnosed, non-metastatic patients whose primary cancer treatment is surgery. Participants will go through initial screening and will be sent an online participant information sheet and consent form. Once consent form is signed, marking enrolment in the study, the second stage of screening will commence. It involves assessing current sleep status (based on diagnostic criteria for acute insomnia) current psychiatric symptoms and review of other relevant medical information (diagnosis of other sleep disorders, other medical and psychiatric disorders). This is to confirm the diagnosis of acute insomnia and establish that there are no medical or psychiatric conditions that might preclude someone from taking part in the study. Once eligibility is ascertained, patients will be randomly assigned to SRT or the SHE control group. The investigators aim to randomise 50 patients (n=25 in each trial arm).

After randomisation to SRT or SHE, patients will be sent an email with a link to complete a baseline (pre-intervention) assessment of sleep, fatigue, and mental health. Patients will also be required to complete the consensus sleep diary and wear an actigraphy device for 7 days prior to commencement of SRT/SHE to record sleep and rest/activity rhythms. After completion of the baseline assessment, patients will either be referred to the research nurse for commencement of the SRT protocol or provided with the SHE resource. At 6 weeks, and 3 months post-randomisation, patients will be requested to complete the same battery of questionnaires as during the baseline assessment. Following completion of the final study assessment (3 months post-randomisation), those randomised to the SHE condition will be offered the opportunity to complete the SRT protocol without the requirement to complete any further assessments.

Interventions: Sleep Restriction Therapy (SRT)

SRT is a manualised, adaptive, behavioural insomnia intervention that is a key active ingredient within multi-component CBT-I. Those randomised to the SRT arm will receive two online sessions supported by two telephone calls over a 4-week intervention phase. SRT will be delivered by trained research nurses.

Sleep Hygiene Education (SHE)

SHE will be delivered via a booklet that provides information about lifestyle changes (e.g., reducing exercise in the evening, light snack before bedtime, reducing caffeine) and changes to the bedroom environment (e.g., dark room, comfortable mattress, optimal room temperature). Patients in the SHE condition will be instructed to implement the SHE advice over a 4-week period.

ELIGIBILITY:
Inclusion Criteria:

Participant is willing and able to give informed consent

Aged 18 years and above

Screen positive for acute insomnia, defined as dissatisfaction with sleep quality or duration, accompanied by other night / daytime symptoms, present for between 2 weeks and 3 months

Newly diagnosed with non-metastatic breast cancer

Primary cancer treatment is surgery

Exclusion Criteria:

* Main study exclusion criteria are limited to conditions contraindicated for SRT or factors that would preclude implementation of SRT.

  1. Pregnancy
  2. Additional sleep disorder diagnosis (e.g., restless legs syndrome, obstructive sleep apnoea, narcolepsy) or screen "positive" for additional sleep disorder at study screening interview
  3. Dementia / Mild Cognitive Impairment
  4. Epilepsy
  5. Psychosis (schizophrenia, bipolar disorder)
  6. Current suicidal ideation with intent or attempted suicide within past 2 months
  7. Night, evening, early morning, or rotating shiftwork
  8. Current / previous psychological treatment for insomnia during the last 12 months
  9. Chemotherapy and / or radiotherapy commenced

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | Screening
  Enrolment logs for all consenting patients. Pre-screen failure logs for patients who meet inclusion criteria but are not enrolled
Retention rates | 3 months post randomisation
  Completion of outcome measures
Intervention fidelity: Therapist adherence | 6 weeks post randomisation
  Independent clinician review of recorded SRT sessions and completion of fidelity rating scale
Intervention fidelity: Patient engagement | During intervention phase
  Intervention attendance logs
  completion of fidelity rating scale
Intervention fidelity: Control group contamination | 6 weeks and 3 months post randomisation
  Client Service Receipt Inventory
Outcome measure completion | Baseline, 6 weeks and 3 months post randomisation
  Completion of study questionnaires
Intervention acceptability | Beginning 8 weeks post-randomisation to approx. 1 year after start of recruitment
  semi-structured interviews with 10 patients from SRT arm, 5 from SHE arm and with 5 members of clinical staff

SECONDARY OUTCOMES:
Improvement in insomnia severity | Baseline, 6 weeks and 3 months post-randomisation
  Insomnia Severity Index (ISI)
Improvement in mental health [depression] | Baseline, 6 weeks and 3 months post-randomisation
  Patient Health Questionnaire 9 (PHQ-9)
Improvement in mental health [anxiety] | Baseline, 6 weeks and 3 months post-randomisation
  Generalised Anxiety Disorders - 7 (GAD-7)
Improvement in rest-activity rhythms [fatigue]Fatigue (FACT-F) | Baseline, 6 weeks and 3 months post-randomisation
  Functional Assessment of Cancer Therapy -
Improvement in rest-activity rhythms | Baseline, throughout the intervention phase, 6 weeks and 3 months post-randomisation
  Actigraphy
Improvement in sleep [estimates of subjective sleep] | Baseline, throughout the intervention phase, 6 weeks and 3 months post-randomisation
  Sleep Diary
Measure of health related quality of life | Baseline, 6 weeks and 3 months post-randomisation
  EQ-5D-5L

REFERENCES:
- [Derived] Fleming L, Zibaite S, Kyle SD, Boyd K, Green V, Mansell J, Elsberger B, Young D. Insomnia prehabilitation in newly diagnosed breast cancer patients: Protocol for a pilot, multicentre, randomised controlled trial comparing nurse delivered sleep restriction therapy to sleep hygiene education (INVEST trial). PLoS One. 2024 Aug 14;19(8):e0305304. doi: 10.1371/journal.pone.0305304. eCollection 2024. PMID 39141622